CLINICAL TRIAL: NCT01924975
Title: Ultrasound-image Guided Versus Traditional Landmark Technique for Saphenous Vein Cannulation in Infants and Small Children
Brief Title: Saphenous Vein Cannulation in Infants and Small Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satoshi Hanada (Other)
Responsible Party: Sponsor-Investigator, Satoshi Hanada, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: V-line study
Record Dates: First submitted 2013-08-14; First posted 2013-08-19 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Saphenous Vein Cannulation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Landmark group (Active Comparator): An operator is not allowed to use an ultrasound. A 22 or 24 G catheter will be advanced blindly toward the expected location of the saphenous vein at the level of the medial malleolus. Once blood appears in the hub, then the catheter will be advanced into the saphenous vein.
  Interventions: Procedure: Saphenous vein cannulation; Device: A 22 or 24 G intravenous catheter
- Ultrasound group (Active Comparator): An operator will identify the saphenous vein by using ultrasound with a linear transducer (L15-7io) in short axis view. A 22 or 24 G catheter will be advanced until the tip of the needle is seen on the ultrasound image. The needle is then advanced until blood appears in the hub. The catheter is then advanced into the saphenous vein.
  Interventions: Procedure: Saphenous vein cannulation; Device: ultrasound with a linear transducer (L15-7io); Device: A 22 or 24 G intravenous catheter

INTERVENTIONS:
Procedure: Saphenous vein cannulation — Intravenous cannulation to saphenous vein
Device: ultrasound with a linear transducer (L15-7io) — Portable, bed-side ultrasound to detect saphenous vein
  Arms: Ultrasound group
Device: A 22 or 24 G intravenous catheter

SUMMARY:
The purpose of this study is to compare the two different saphenous vein cannulation techniques; real-time ultrasound image-guided technique (Ultrasound group) vs. traditional landmark technique (Landmark group).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patient undergoing scheduled surgery which requires venous cannulation.
2. Term neonates and children < 4 years old weighing >/= 3 kg

Exclusion Criteria:

1. Patient with visible saphenous vein
2. Patient with no detectable saphenous vein under ultrasound
3. Patient with a skin wound or infection around puncture site
4. Patient with recent venous puncture at the puncture site (less than 1 month)
5. Patient with thrombus in saphenous vein or hematoma formation around the vein detected by ultrasound.
6. Patient with any emergency surgery

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Hanada, MD, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Triffterer L, Marhofer P, Willschke H, Machata AM, Reichel G, Benkoe T, Kettner SC. Ultrasound-guided cannulation of the great saphenous vein at the ankle in infants. Br J Anaesth. 2012 Feb;108(2):290-4. doi: 10.1093/bja/aer334. Epub 2011 Oct 27. PMID 22037223
- [Background] Riera A, Langhan M, Northrup V, Santucci K, Chen L. Remember the saphenous: ultrasound evaluation and intravenous site selection of peripheral veins in young children. Pediatr Emerg Care. 2011 Dec;27(12):1121-5. doi: 10.1097/PEC.0b013e31823ab926. PMID 22134232
- [Background] Joshi M, Wilson G, Engelhardt T. Comparison of landmark technique and ultrasound guidance for localisation of long saphenous vein in infants and children. Emerg Med J. 2010 Jun;27(6):443-5. doi: 10.1136/emj.2008.069310. PMID 20562139

RESULTS

PARTICIPANT FLOW:
Groups:
- Landmark Group: An operator is not allowed to use an ultrasound. A 22 or 24 G catheter will be advanced blindly toward the expected location of the saphenous vein at the level of the medial malleolus. Once blood appears in the hub, then the catheter will be advanced into the saphenous vein.
  Saphenous vein cannulation: Intravenous cannulation to saphenous vein
  A 22 or 24 G intravenous catheter
- Ultrasound Group: An operator will identify the saphenous vein by using ultrasound with a linear transducer (L15-7io) in short axis view. A 22 or 24 G catheter will be advanced until the tip of the needle is seen on the ultrasound image. The needle is then advanced until blood appears in the hub. The catheter is then advanced into the saphenous vein.
  Saphenous vein cannulation: Intravenous cannulation to saphenous vein
  ultrasound with a linear transducer (L15-7io): Portable, bed-side ultrasound to detect saphenous vein
  A 22 or 24 G intravenous catheter
Period: Overall Study
Arm/Group | Landmark Group | Ultrasound Group
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Landmark Group | Ultrasound Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 12 [6 to 29] | 8 [4 to 26] | 11 [5 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 27 | 35 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Attempt Success of Saphenous Vein Cannulation
Time Frame: 10 minutes
Measure: Number; unit: percent of participants
Arm/Group | Landmark Group | Ultrasound Group
Number analyzed (Participants) | 51 | 51
percent of participants | 51.0 | 90.2

2. Secondary Outcome: Percentage of Participants With Success of Saphenous Vein Cannulation Within 3 Attempts of Needle Insertion, or a 10 Minute Time Period.
Time Frame: 10 minutes
Measure: Number; unit: percent of participants
Arm/Group | Landmark Group | Ultrasound Group
Number analyzed (Participants) | 51 | 51
percent of participants | 62.8 | 92.2

3. Secondary Outcome: Time Required for Overall Successful Venous Cannulation.
Time Frame: 10 minutes
Population: Includes only those participants for which successful cannulation was achieved.
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Landmark Group | Ultrasound Group
Number analyzed (Participants) | 32 | 47
Seconds | 235 [179 to 300] | 151 [112 to 246]

ADVERSE EVENTS:
Arm/Group | Landmark Group | Ultrasound Group
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No